CLINICAL TRIAL: NCT03810196
Title: CD45RA Depleted Peripheral Stem Cell Addback for Patients At Risk for Viral or Fungal Infections Post TCRαβ/CD19 Depleted Hematopoietic Stem Cell Transplant
Brief Title: CD45RA Depleted Peripheral Stem Cell Addback for Viral or Fungal Infections Post TCRαβ/CD19 Depleted HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Olson, Medical Director, Hematopoietic Stem Cell Transplantation (HSCT) Program, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-015286
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Acute Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Acute Lymphoblastic Leukemia; Mixed Lineage Leukemia; Lymphoblastic Lymphoma; Burkitt Lymphoma; Juvenile Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia, Myelomonocytic, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TBI regimen (Other): Standard of care myeloablative regimens will be used based on disease type and clinical status at time of transplant. Patients with acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma will receive total body irradiation (TBI) regimen (thiotepa, cyclophosphamide, TBI).
  Interventions: Device: CliniMACS Cell Processing System for TCRαβ + T Cell and CD45RA Depleted Peripheral Stem Cell Addback
- TBI or busulfan regimen (Other): Standard of care myeloablative regimens will be used based on disease type and clinical status at time of transplant. Patients not diagnosed with ALL or lymphoblastic lymphoma may receive either total body irradiation (TBI) regimen (thiotepa, cyclophosphamide, TBI) or busulfan containing regimen (thiotepa, cyclophosphamide, busulfan).
  Interventions: Device: CliniMACS Cell Processing System for TCRαβ + T Cell and CD45RA Depleted Peripheral Stem Cell Addback

INTERVENTIONS:
Device: CliniMACS Cell Processing System for TCRαβ + T Cell and CD45RA Depleted Peripheral Stem Cell Addback — Peripheral stem cell (PSC) product will be processed using the CliniMACS device for TCRαβ and T cell depletion. Approximately 10% of the PSCs will undergo CD45RA depletion and cryopreservation. Patients will receive CD45RA depleted infusion after the TCRab PSCT.

SUMMARY:
The major morbidities of allogeneic hematopoietic stem cell transplant with non-human leukocyte antigen (HLA) matched siblings are graft vs host disease (GVHD) and life threatening infections. T depletion of the donor hematopoietic stem cell graft is effective in preventing GVHD, but immune reconstitution is slow, increasing the risk of infections. An addback of donor CD45RA (naive T cells) depleted cells may improve immune reconstitution and help decrease the risk of infections.

DETAILED DESCRIPTION:
The risk of severe graft versus host disease (GVHD) is increased with the use of unrelated and partially matched related donors. T cell depletion reduces the risk of severe GVHD, but immune reconstitution is delayed. Important memory T cells that may protect patients from fungal and viral infections are also removed in the T depletion process. CD45RA depletion has been studied both as a single step to reduce the risk of GVHD, and also, in conjunction with αβTCR depleted hematopoietic stem cell grafts to accelerate immune reconstitution. This is a single institutional pilot trial of this T cell depletion technique. Patients with acute leukemias at high risk for relapse are eligible to participate. Patients will be given CD45RA depleted donor peripheral stem cells (PSCs) following T depleted hematopoietic stem cell transplant (HSCT). A short course of GVHD prophylaxis will be used after CD45RA depletion.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients <25 years.
2. First allogeneic HSCT only.
3. Disease eligibility: Acute leukemias at high risk for relapse including positive minimal residual disease at end consolidation, high risk cytogenetics, or relapse. Hematologic malignancies including: acute myeloid leukemia, myelodysplastic syndromes, acute lymphoblastic leukemia, mixed lineage or bi-phenotypic leukemia, lymphoblastic or Burkitts, juvenile myelomonocytic leukemia
4. Evaluation of organ and infectious status as per our Bone Marrow Transplant standard operating procedure (BMT SOP).
5. Signed consent by parent/guardian or able to give consent if >18 years.

Exclusion Criteria:

1. Patients who do not meet institutional disease, organ or infectious criteria
2. No suitable donor available for mobilized peripheral stem cells
3. Patients with genetic disorders including Fanconi anemia, Kostmann syndrome, dyskeratosis congenital or other DNA repair defects.
4. Patients with Hodgkin lymphoma or non-Burkitts, non-lymphoblastic lymphoma
5. Pregnant Participants

Donor selection and eligibility

1. Unrelated donor meets National Marrow Donor Program criteria for donation
2. HLA testing/matching
3. Donor must be willing to undergo granulocyte colony stimulating factor (GCSF) mobilization and peripheral blood stem cell collection

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute graft vs. host disease (GVHD) | Up to 100 days post-transplantation
  Incidence of acute graft vs. host disease (GVHD) (reaction of donor immune cells against host tissues)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No